CLINICAL TRIAL: NCT05369000
Title: A Phase 1 Open-label Trial to Evaluate the Safety, Tolerability, PK, PD, Immunogenicity, and Antitumor Activity of LAVA-1207, a PSMA-targeting Bispecific γδ-T Cell Engager, Alone or With Low Dose Interleukin-2 or Pembrolizumab, in Patients With Therapy Refractory mCRPC
Brief Title: Trial of LAVA-1207 in Patients With Therapy Refractory Metastatic Castration Resistant Prostate Cancer (mCRPC) Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was intended to be a Phase 1/2 trial (but the trial never moved forward to Phase 2).
Sponsor: Lava Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LAVA1207-001/LAVA1207-002; 2021-001789-39 (EudraCT Number); KEYNOTE-F73 (Other: Merck Sharp & Dohme, LLC)
Record Dates: First submitted 2022-04-29; First posted 2022-05-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: prostate cancer; PSMA; mCRPC; Phase 1 dose escalation; Phase 1 safety; Phase 2 safety; open-label
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- LAVA-1207 (Experimental): LAVA-1207
  Interventions: Biological: LAVA-1207
- LAVA-1207 with Low-Dose Subcutaneous IL-2 (LDSC IL-2) (Experimental): LAVA-1207 with Low-Dose Subcutaneous IL-2 (LDSC IL-2)
  Interventions: Biological: LAVA-1207
- LAVA-1207 plus Pembrolizumab (Experimental): LAVA-1207 plus Pembrolizumab
  Interventions: Biological: LAVA-1207; Biological: LAVA-1207 plus Pembrolizumab

INTERVENTIONS:
Biological: LAVA-1207 — In part 1 & part 2
  • LAVA-1207 will be administered via intravenous infusion.
Biological: LAVA-1207 plus Pembrolizumab — Pembrolizumab will be administered via intravenous infusion
  Arms: LAVA-1207 plus Pembrolizumab

SUMMARY:
This is a phase 1, first-in-human study to evaluate Safety, Tolerability, PK, PD, Immunogenicity, and Antitumor Activity of LAVA-1207 alone or with low dose interleukin-2 or Pembrolizumab, in patients with therapy refractory metastatic castration resistant prostate cancer.

DETAILED DESCRIPTION:
This trial is an open-label Phase 1 dose escalation trial with an expansion cohort to investigate the safety and tolerability of LAVA-1207 alone or with low dose interleukin-2 or Pembrolizumab, in patients with therapy refractory mCRPC.

The trial was intended to be a Phase 1/2 trial (but the trial never moved forward to Phase 2).

ELIGIBILITY:
INCLUSION CRITERIA (for patients receiving LAVA-1207 +/- LDSC IL-2):

Patients are eligible to be included in the arm only if all of the following criteria apply:

1. Patient must be 18 years of age inclusive or above, at the time of signing the informed consent.
2. Male patient with mCRPC as defined by PCWG3 criteria (histologically confirmed adenocarcinoma; adenocarcinoma with ≤10% small-cell or neuroendocrine features is allowed). Brain metastases are allowed as long as the patient's symptoms are well controlled.
3. Patient should have failed at least 1 line of taxane-based chemotherapy or is deemed medically unsuitable to be treated with a taxane regimen.
4. Patient should have received a 2nd generation or later androgen receptor targeted therapy/ androgen biosynthesis inhibitor (e.g., abiraterone,enzalutamide, and/or apalutamide). Progression on novel antiandrogen therapy may have occurred in the non-mCRPC setting.
5. Patient is unlikely to tolerate or derive clinically meaningful benefit from other available therapy.
6. Patient for which any drug-related toxicity adverse effects of any prior cancer therapy have resolved to Grade 1 or less according to CTCAE version 5.0 or to baseline severity level (except for alopecia and peripheral neuropathy).
7. Patients with evidence of progressive disease, defined as 1 or more of the following criteria:

   1. PSA level ≥1 ng/mL that has increased on at least 2 successive occasions at least 1 week apart.
   2. Computed tomography (CT) or magnetic resonance imaging (MRI) scan: nodal or visceral progression as defined by RECIST 1.1.
   3. Bone scintigraphy: appearance of 2 or more new metastatic lesions.
8. Patient should have undergone bilateral orchiectomy or should be on continuous androgen-deprivation therapy (ADT) with a gonadotropin-releasing hormone agonist or antagonist (surgical or medical castration).
9. Total serum testosterone ≤ 50 ng/dL or 1.73 nmol/L.
10. Evaluable (measurable or non-measurable) disease for prostate cancer.
11. Predicted life-expectancy of ≥ 6 months.
12. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
13. Adequate renal function (estimated glomerular filtration rate [eGFR] per local laboratory > 40 mL/min/1.73m2), hepatic (bilirubin ≤ 2 times upper limit of normal [ULN], aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≤3.0 times ULN). In case of liver metastases, AST, and ALT ≤ 5.0 times ULN is allowed. Adequate hematological function (neutrophils > 1 x 109/L, platelet count > 75 x 109/L, Hb>9g/dL) with no prior transfusions within 2 weeks.
14. Males who are:

    1. Surgically sterile (bilateral orchiectomy, vasectomy).
    2. Compliant with an effective contraceptive regimen (i.e. use of male condom with female partner and assuring use of an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a woman of childbearing potential who is not currently pregnant) following from signing of the informed consent form [ICF] through 90 days after the last IMP administration. Abstinence is not considered an adequate contraceptive regimen.
    3. Refraining from donating sperm following the signing of the ICF through 90 days after the last IMP administration.
15. Capable of giving signed and dated informed consent prior to initiation of any trial-related procedures that are not considered Standard of Care which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

INCLUSION CRITERIA (for LAVA-1207 plus pembrolizumab arm):

Patients are eligible to be included in the arm only if all of the following criteria apply:

1. Patient must be 18 years of age inclusive or above, at the time of signing the informed consent.
2. Male patient with mCRPC as defined by PCWG3 criteria (histologically confirmed adenocarcinoma; adenocarcinoma with ≤10% small-cell or neuroendocrine features is allowed). Brain metastases are allowed as long as the patient's symptoms are well controlled, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
3. Patient should have failed at least 1 line of taxane-based chemotherapy or is deemed medically unsuitable to be treated with a taxane regimen.
4. Patient should have received a 2nd generation or later androgen receptor targeted therapy/androgen biosynthesis inhibitor (e.g., abiraterone, enzalutamide, and/or apalutamide). Progression on novel anti-androgen therapy may have occurred in the non-mCRPC setting.
5. Patient is unlikely to tolerate or derive clinically meaningful benefit from other available therapy.
6. Patient for which any drug related toxicity or adverse effects of any prior cancer therapy should have resolved to Grade 1 or less according to CTCAE version 5.0 or to baseline severity level (except alopecia and peripheral neuropathy).
7. Patient has evidence of progressive disease, defined as 1 or more criteria:

   1. PSA level ≥1 ng/mL that has increased on at least 2 successive occasions at least 1 week apart.
   2. CT or MRI scan: nodal or visceral progression as defined by RECIST 1.1.
   3. Bone scintigraphy: appearance of 2 or more new metastatic lesions.
8. Patient should have undergone bilateral orchiectomy or should be on continuous ADT with a gonadotropin-releasing hormone agonist or antagonist (surgical or medical castration).
9. Total serum testosterone ≤ 50 ng/dL or 1.73 nmol/L.
10. Evaluable (measurable or non-measurable) disease for prostate cancer.
11. Predicted life-expectancy of ≥ 6 months.
12. ECOG performance status of 0 or 1.
13. Adequate renal function (eGFR per local laboratory > 40 mL/min/1.73m2), hepatic (bilirubin < 1.5 times ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5 × ULN, AST and ALT <2.5 times ULN). In case of liver metastases, AST, and ALT < 5.0 times ULN is allowed. Adequate hematological function (neutrophils > 1.5 x109/L, platelet count > 100x109/L, Hb>9g/dL or 5.6 mmol/L, with no prior transfusions within two weeks).
14. Males who are:

    1. Surgically sterile (bilateral orchiectomy, vasectomy).
    2. Compliant with an effective contraceptive regimen (i.e., use of male condom with female partner and assuring use of an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a woman of childbearing potential who is not currently pregnant following from signing of the ICF through 90 days after the last IMP administration). Abstinence is not considered an adequate contraceptive regimen.
    3. Refraining from donating sperm following the signing of the ICF through 90 days after the last IMP administration.
15. Capable of giving signed and dated informed consent prior to initiation of any trial-related procedures that are not considered Standard of Care which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

EXCLUSION CRITERIA (for patients receiving LAVA-1207 +/- LDSC IL-2):

Patients are excluded from the trial if any of the following criteria apply:

1. Other malignancies within the last 2 years except adequately treated carcinoma in situ, basal or squamous cell skin carcinoma.
2. Uncontrolled or severe intercurrent medical condition.
3. Positive serological testing for human immunodeficiency virus (HIV) antibody.
4. Positive serological hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (anti-HBc) negative, and hepatitis C virus (HCV) antibody. Patients who are positive for anti-HBc or hepatitis C antibody may be included if they have a negative polymerase chain reaction (PCR) within 6 weeks prior to initial IMP administration. Those who are PCR positive will be excluded.
5. Patient has any active, uncontrolled, or suspected infection.
6. Known clinically relevant immunodeficiency disorders.
7. A significant history of renal, neurologic, psychiatric, pulmonary, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the investigator would adversely affect participation in this trial.
8. Unstable cardiovascular function defined as: (a) symptomatic ischemia, or (b) uncontrolled clinically significant conduction abnormalities (i.e. ventricular tachycardia on antiarrhythmic agents are excluded; 1st degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block is not excluded), or (c) congestive heart failure New York Heart Association Class ≥ 3, or (d) myocardial infarction within 3 months.
9. Previous treatment with antitumor therapies within 2 weeks prior to initial IMP for radiotherapy and androgen receptor targeted therapy/androgen biosynthesis inhibitor, and within 4 weeks for systemic chemotherapy or targeted immunotherapy.
10. Previous treatment with live or live attenuated vaccines within 2 weeks prior to initial IMP administration. New types of vaccines need to be evaluated as to their mode of action.
11. Treatment with other investigational agents in the 4 weeks prior to initial IMP administration.
12. Major surgery within 4 weeks prior to initial IMP administration.
13. Hypersensitivity to any of the excipients present in LAVA-1207 or IL-2 (if applicable).
14. Previous treatment with any systemic immunosuppressant within 4 weeks prior to initial IMP administration, with the exception of systemic corticosteroid use up to oral dose of 10 mg prednisone daily (or equivalent for other steroids).
15. Previous treatment with an aminobisphosphonate IV (e.g., ibandronate, pamidronate, zoledronate etc.) within 12 months prior to initial IMP.
16. Known ongoing drug and alcohol abuse in the opinion of the investigator.

EXCLUSION CRITERIA (for LAVA-1207 plus pembrolizumab arm):

Patients are excluded from the arm if any of the following criteria apply:

1. Other malignancies within the last 2 years except adequately treated carcinoma in situ, basal or squamous cell skin carcinoma.
2. Seropositive for and with evidence of active viral infection with hepatitis B virus (HBV). Patients who are HBsAg negative and HBV viral DNA negative are eligible. Patients who had HBV but have received an antiviral treatment and show non-detectable viral DNA for 6 months are eligible. Patients who are seropositive because of HBV vaccine are eligible.
3. Seropositive for and with active viral infection with hepatitis C virus (HCV). Patients who had HCV but have received an antiviral treatment and show no detectable HCV viral DNA for 6 months are eligible.
4. History of allogenic tissue or solid organ transplant.
5. Positive serological testing for HIV.
6. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
7. Hypersensitivity to any of the excipients present in LAVA-1207.
8. Active infection requiring systemic therapy.
9. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
12. Has received prior therapy with an anti-programmed cell death 1 (PD 1), anti-programmed cell death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher immune related AE (irAE).
13. A significant history of renal, neurologic, psychiatric, pulmonary, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the investigator would adversely affect participation in this trial.
14. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
15. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks (could consider shorter interval for kinase inhibitors or other short half-life drugs) prior to treatment. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs ≤Grade 2 requiring treatment or hormone replacement may be eligible. Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
16. Has received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis. Note: Participants must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
17. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Note: Administration of killed vaccines are allowed.
18. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
19. Major surgery within 4 weeks prior to initial IMP administration.
20. Previous treatment with an aminobisphosphonate IV (e.g., ibandronate, pamidronate, zoledronate etc.) within 12 months prior to initial IMP.
21. Known ongoing drug and alcohol abuse in the opinion of the investigator.
22. Patients will be unlikely to tolerate or derive clinically meaningful benefit from other available therapy.
23. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
24. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 96 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Part 1 & Part 2: Frequency and severity of AEs | Approximately 24 months
  Frequency and severity of Adverse Events using the Common Terminology Criteria and grading for Adverse Events and grading for CRS
Part 1: Frequency and type of DLT | First 28 days of treatment
  DLT is defined as an adverse event that is unrelated to disease progression, intercurrent illness, or concomitant medications and is occurring during the first 28 days of treatment.illness, or concomitant medications and is occurring during the first 28 days of treatment.

SECONDARY OUTCOMES:
Part 1 & Part 2: Number of participants with an antitumor response | Approximately 24 months
  According to immune Response Evaluation Criteria in Solid Tumors (RECIST and iRECIST) in patients with measurable disease.
Part 1 & Part 2: Pharmacokinetic of LAVA-1207, area under the concentration versus time curve (AUC) | Approximately 6 months
  Area under the plasma concentration versus time curve (AUC) of LAVA-1207 will be assessed in all patients
Part 1 & Part 2: Incidence and prevalence of anti-LAVA-1207 antibodies | Approximately 6 months
  Development of antibodies (anti-drug antibodies) to LAVA-1207 will be evaluated
Part 1 & Part 2: Biomarkers, binding of LAVA-1207 to Vγ9Vδ2-T cells | Approximately 24 months
  Binding of LAVA-1207 to Vγ9Vδ2-T cells will be measured in whole blood

OTHER OUTCOMES:
Exploratory Objective | Approximately 24 months
  To evaluate the effect of study treatment on circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Management, Study Director — Lava Therapeutics
Locations (12):
- United States (6):
  - UCSF Medical Center at Parnassus, San Francisco, California
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Duke University Medical Center - Duke Cancer Center, Durham, North Carolina
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
- Netherlands (3):
  - Radboud Universiteit - Radboud Universitair Medisch Centrum (Radboudumc), Nijmegen, Gelderland
  - Erasmus MC (Erasmus Universitair Medisch Centrum Rotterdam), Rotterdam, South Holland
  - Amsterdam UMC - VU Medisch Centrum (VUmc), Amsterdam
- Spain (3):
  - ICO Hospitalet (Hospital Duran i Reynals), Barcelona
  - Hospital Universitartio 12 De Octubre, Madrid
  - Centro Integral Oncologico Clara Campal (HM CIOCC), Madrid

IPD SHARING:
Plan to Share IPD: No